CLINICAL TRIAL: NCT03956329
Title: Enhancing Influenza Vaccination by Optimising Mood in Older Adults: a Randomised Controlled Clinical Trial
Brief Title: Flu and Mood in Older Adults
Acronym: For-ME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Public Health England (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 19004
Record Dates: First submitted 2019-04-30; First posted 2019-05-20 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Vaccination; Infection
Keywords: Positive Affect; Influenza Vaccination; Positive Mood; Vaccination; Randomised Control Trial
MeSH Terms: conditions — Infections; Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Note: Blinding not possible for usual care group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care, control arm (No Intervention): Usual care in which participants will not see a video intervention. This group will attend their influenza vaccination appointment as usual, without intervention. Participants will receive Northern Hemisphere Influenza Vaccine 2019/20 (Delivered as part of Standard Care).
- Standardised Digital Intervention (Experimental): Video intervention designed to induce an increase in positive mood in older adults. Includes comedy clips, uplifting music and positive imagery. Intervention approximately 15-20 minutes in length. Following intervention, participants will receive the Northern Hemisphere Influenza Vaccine 2019/20 (Delivered as part of Standard Care).
  Interventions: Other: Standardised Digital Intervention
- Individualised Digital Intervention (Experimental): Similar to the standardised digital intervention, however participants will be able to individualise the intervention by choosing video clips from a limited menu of choices. Intervention approximately 15-20 minutes in length. Following intervention, participants will receive the Northern Hemisphere Influenza Vaccine 2019/20 (Delivered as part of Standard Care).
  Interventions: Other: Individualised Digital Intervention

INTERVENTIONS:
Other: Standardised Digital Intervention — Video intervention designed to induce an increase in positive mood in older adults. Includes comedy clips, uplifting music and positive imagery. Intervention approximately 15-20 minutes in length. This includes 3 short comedy clips (fork handles sketch, the two Ronnie's; A room with a view - faulty towers; Tim Vine Live stand-up extract), uplifting music (Jailhouse Rock - Elvis Presley; Happy Together - The Turtles), jokes and positive imagery. The content of the intervention has been informed by patient and public involvement, focus groups with older adults, and pilot testing.
  Arms: Standardised Digital Intervention
Other: Individualised Digital Intervention — Similar to the standardised digital intervention, however, participants will be able to individualise the intervention by choosing video clips from a limited menu of choices. Intervention approximately 15-20 minutes in length. The 4 categories include stand-up comedy (Michael McIntyre, Tim Vine and Victoria Wood), sit-com (Fawlty Towers, Only Fools and Horses and Two Ronnies), music (Elvis Presley, Last Night at the Proms, Roy Orbison) and variety (Britain's Got Talent, Strictly Come Dancing, Terry Wogan). Participants are able to select 3 of the videos, which are roughly 5 minutes in length, to reach a total of 15-20 minutes of content.
  Arms: Individualised Digital Intervention

SUMMARY:
Randomised control trial comparing the effects of a standardised and individualised positive affect digital intervention versus usual care on mood and antibody responses to influenza vaccination in older adults.

DETAILED DESCRIPTION:
Infectious diseases are important causes of morbidity and mortality worldwide, and vaccinations are vital to reducing the risk of disease. Vaccine efficacy, however, is dependent on the immune system's ability to respond to vaccination antigens. Influenza vaccines play an important role in combating influenza. However, some populations, such as older adults, respond poorly to vaccination due to their compromised immune systems, with efficacy at 17-53% (compared to 70-90% in young adults).

Behavioural and psychological influences have been shown to alter immune responses. An observational study looking into behavioural and psychological effects, which have been identified as immune modulators (stress, physical activity, nutrition, mood and sleep) found greater positive mood on the day of vaccination predicted significantly greater antibody responses to influenza vaccination. Following this, a feasibility study carried out on 110 older adults demonstrated the ability to enhance positive mood prior to influenza vaccination using a brief digital intervention.

The clinical trial will be the next phase of this research, where the cohort will consist of 650 participants, aged over 65 years, who will receive the quadrivalent, cell-grown influenza vaccination, immediately after one of three conditions. These conditions include: the control arm of usual participant care for vaccination; participants watching a 15-minute digital intervention via a tablet that does not allow content selection; and a personalised digital intervention that allows for participant selection of content they would like to view for 15 minutes. The purpose of these digital interventions is to enhance positive mood of patients prior to vaccination.

The primary aim of this trial is to explore which of two brief interventions has the largest effect on positive mood, compared with usual care. The secondary aim is to measure vaccine specific antibody responses, with the hypothesis that individuals with enhanced positive mood will present larger vaccine specific antibody responses.

This trial will also allow data collection on exploring recruitment, attrition, intervention engagement, and practicality of collecting clinical data available through electronic records and self-report measures to inform the design of a future definitive trial.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females aged 65-85 years (inclusive)
* Received influenza vaccination for the 2018/19 season
* Eligible to receive 2019/20 influenza vaccination as part of usual care
* Ability to give informed consent

Exclusion Criteria:

* Males and Females aged less than 65 or over 85 years (exclusive)
* Did not receive influenza vaccination for the 2018/19 season
* Ineligible to receive 2019/20 influenza vaccination as part of usual care
* Unable to provide informed consent
* Deemed by health care provider to be:
* Too physically frail to participate
* Diagnosed with dementia or other cognitive condition which would make participation difficult
* Insufficient command of English language
* Influenza vaccination contraindicated
* Sufficiently impaired of hearing or vision that exposure to the intervention video content as intended would be compromised
* Those for whom the collection of blood samples is contraindicated
* Those who have participated previously in the pilot study (NCT03144518).

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 654 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Self-Reported Mood- Affective Slider | Baseline, immediately post- intervention (15- 20 minutes post baseline)
  Self-reported mood will be measured using three validated patient-reported outcome measures to determine changes in mood from before to after usual care/ intervention arms. One of the three outcome measures includes the Affective Slider (AS), which is a slider scale that is measures a single value on a continuous normalised scale ranging from 0-1, with a central, default thumb position value equal to 0.5, where 0 is low and 1 is high.
Self-Reported Mood- Scale of Positive and Negative Experience | Baseline, immediately post- intervention (15- 20 minutes post baseline)
  The second outcome measure of changes in mood will be the Scale of Positive and Negative Experience (SPANE), where participants rate 12 emotion words from 1 to 5, where 1 is Not at all and 5 is Very. The overall affect is then determined using these scores and can also be divided out into positive and negative feelings scales.
Self-Reported Mood- Happy-Sad and Alert-Sleepy Dynamic Visual Analogue Mood Scales | Baseline, immediately post- intervention (15- 20 minutes post baseline)
  The third and final measure of changes in mood will be the Happy-Sad and Alert-Sleepy Dynamic Visual Analogue Mood Scales (DVAMS), which is a morphing image scale that is gender specific and changes when the participant moves the slider scale. The scale ranges from 0 to 100, where 0 is low and 100 is high. The central, default thumb position value is 50.

SECONDARY OUTCOMES:
Influenza vaccination-specific antibody responses- Haemagglutination inhibition assay | Baseline, 4 weeks post-vaccination
  Antibody levels specific to antigens contained in the influenza vaccination will be assessed in sera taken immediately prior to vaccination and at 4 weeks post-vaccination. This will be assessed using the haemagglutination inhibition (HAI) assay that allows for the determination of the quantity of influenza virus present based of HAI units by carrying out serial dilutions. A larger number of HAI units equates to a high quantity of influenza virus.
Influenza vaccination-specific antibody responses- IgG-specific enzyme-linked immunosorbent assay | Baseline, 4 weeks post-vaccination
  The concentration of influenza specific antibody will be measured using a IgG- specific enzyme linked immunosorbent assay (ELISA).
Number of participants who experience flu-like symptoms and self care | 6 months
  Participants who experience cold and flu-like symptoms will a complete flu-like symptoms diary and self-care behaviours for occasions of flu-like illnesses during the 6 months post-vaccination.
Number of participants who do not follow up with trial procedures- Attrition | Baseline, immediately post- intervention, 4 weeks post-vaccination, 6 months post-vaccination
  Loss to follow-up will be noted for participants who do not complete the intervention, do not attend the post-vaccination follow-up, and who do not return flu-like symptom diaries at 6 months post-vaccination.
Recruitment | From the time of recruitment to the start of the Randomised Control Trial
  The number and proportion of participants who consent to participate in the trial from the total number of the population approached.

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Vedhara, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ayling K, Fairclough L, Tighe P, Todd I, Halliday V, Garibaldi J, Royal S, Hamed A, Buchanan H, Vedhara K. Positive mood on the day of influenza vaccination predicts vaccine effectiveness: A prospective observational cohort study. Brain Behav Immun. 2018 Jan;67:314-323. doi: 10.1016/j.bbi.2017.09.008. Epub 2017 Sep 18. PMID 28923405
- [Background] Andre FE, Booy R, Bock HL, Clemens J, Datta SK, John TJ, Lee BW, Lolekha S, Peltola H, Ruff TA, Santosham M, Schmitt HJ. Vaccination greatly reduces disease, disability, death and inequity worldwide. Bull World Health Organ. 2008 Feb;86(2):140-6. doi: 10.2471/blt.07.040089. PMID 18297169
- [Background] Goodwin K, Viboud C, Simonsen L. Antibody response to influenza vaccination in the elderly: a quantitative review. Vaccine. 2006 Feb 20;24(8):1159-69. doi: 10.1016/j.vaccine.2005.08.105. Epub 2005 Sep 19. PMID 16213065
- [Background] Moynihan JA, Larson MR, Treanor J, Duberstein PR, Power A, Shore B, Ader R. Psychosocial factors and the response to influenza vaccination in older adults. Psychosom Med. 2004 Nov-Dec;66(6):950-3. doi: 10.1097/01.psy.0000140001.49208.2d. PMID 15564363
- [Background] Betella A, Verschure PF. The Affective Slider: A Digital Self-Assessment Scale for the Measurement of Human Emotions. PLoS One. 2016 Feb 5;11(2):e0148037. doi: 10.1371/journal.pone.0148037. eCollection 2016. PMID 26849361
- [Background] Barrows PD, Thomas SA. Assessment of mood in aphasia following stroke: validation of the Dynamic Visual Analogue Mood Scales (D-VAMS). Clin Rehabil. 2018 Jan;32(1):94-102. doi: 10.1177/0269215517714590. Epub 2017 Jun 27. PMID 28653547
- [Derived] Ayling K, Brown M, Carlisle S, Bennett R, Buchanan H, Dumbleton J, Hawkey C, Hoschler K, Jack RH, Nguyen-Van-Tam J, Royal S, Turner D, Zambon M, Fairclough L, Vedhara K. Optimizing mood prior to influenza vaccination in older adults: A three-arm randomized controlled trial. Health Psychol. 2024 Feb;43(2):77-88. doi: 10.1037/hea0001267. Epub 2023 Dec 7. PMID 38059932